CLINICAL TRIAL: NCT06189820
Title: Role of the Fibroblast Activation Protein (FAP) as Biomarker of Fibrotic Lung Diseases
Acronym: FAPIPET
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: P2022/587
Record Dates: First submitted 2023-11-22; First posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-11

CONDITIONS: Pulmonary Fibrosis; Lung Fibrosis; Idiopathic Pulmonary Fibrosis; FAP
Keywords: Pulmonary fibrosis; FAP
MeSH Terms: conditions — Pulmonary Fibrosis; Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: FAPI PET/CT — In the department of Nuclear Medicine:
  * Installation in a relax chair after weight and height control
  * Placement of a venous line in the upper limb after which an infusion of 500ml of 0.9% NaCl is started.
  * Intravenous injection of 3 MBq/kg (max 300 MBq) of 18F- FAPI 74 or of 2 MBq/kg 68Ga-FAPI46

SUMMARY:
To evaluate the effect of an anti-fibrotic treatment initiation on the fibrotic activity as assessed by FAPI PET/CT.

DETAILED DESCRIPTION:
To evaluate the use of the fibroblast activation protein (FAP) as a biomarker of fibrotic lung disease (idiopathic pulmonary fibrosis (IPF) and non-IPF ILDs). The study will include both analysis of FAP expression in samples stored in the biobank of the department of Pneumology (BAL, blood, induced sputum and EBC) (cohort A) and lung FAPI uptake on PET/CT scans performed at the department of Nuclear Medicine:

* before and after the initiation of an antifibrotic therapy (IPF or PPF) (cohort B)
* before and after the initiation of corticosteroid therapy in case of an acute exacerbation of ILD (cohort C)
* before and after the initiation of an immunosuppressive drug in the context of non-IPF pulmonary fibrosis (cohort D).
* before lung transplantation, surgery or biopsy to correlate with FAP expression determined by immunohistochemical analysis (IHC) (cohort E).

ELIGIBILITY:
Inclusion Criteria:

* Adults patients with a fibrotic lung disease (idiopathic pulmonary fibrosis (IPF) or non-IPF fibrotic ILD) as defined according to the 2022 ATS/ERS/JRS/ALAT Clinical Practice Guidelines

Exclusion Criteria:

* Pregnant or nursing patients
* Patients with another significant medical condition which, in the investigator's opinion, may interfere with the completion of the study.
* Patients with an active lung neoplasm or any active neoplasm for blood samples

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-03-09 (Actual); Primary Completion 2027-03-09 (Estimated); Study Completion 2027-03-09 (Estimated)

PRIMARY OUTCOMES:
FAPI uptake on PET/CT | From date of inclusion till date of the second FAPI PET/CT (after 3 months)
  Decrease in lung FAPI uptake after the initiation of treatment, measured with the following PET parameters: SUVmax, SUVmean and Total lesion fapi uptake (TLA) in the lungs of the patients

SECONDARY OUTCOMES:
Correlation between lung FAP expression and clinical evolution | From date of inclusion for a period of 2 years
  Correlation between lung FAP expression (as assessed on blood/BAL or on FAPI PET/CT) and the clinical evolution based on the analysis of the slope of FVC decreased, absolute and relative changes in FVC at 12 months, time to progression/death or lung transplantation, time to first acute exacerbation
Comparison of different FAPi tracers | From date of inclusion till the second FAPi PET/CT (maximum period of 4 weeks)
  Comparison of PET parameters on 68Ga-FAPI and 18F-FAPI images (SUVmax, SUVmean) in lungs
Comparison of different FAPi tracers | From date of inclusion till the second FAPi PET/CT (maximum period of 4 weeks)
  Comparison of PET parameters of 68Ga-FAPI and 18F-FAPI images (SUVmax, SUVmean) in blood pool
Correlation between lung FAPI uptake and corresponding FAP assessment in blood and BAL samples. | From date of inclusion till last BAL sample taken, up to a maximum period of 2 years follow-up
  Correlation between lung FAPI uptake on the PET images (SUVmean, SUVmax, TLA) and corresponding quantitative FAP assessment in blood and BAL samples.
Correlation between lung FAPI uptake and immunohistological evaluation of the FAP expression on lung samples (after lung transplantation, surgical lung biopsy or cryobiopsy) | From date of inclusion until surgery, for a maximum period of 2 years
  Correlation between lung FAPI uptake on the PET images (SUVmean, SUVmax, TLA) and immunohistological evaluation of the FAP expression on lung samples (after lung transplantation, surgical lung biopsy or cryobiopsy)

CONTACTS AND LOCATIONS:
Locations (1):
- Medecine, Brussels, Belgium